CLINICAL TRIAL: NCT04047875
Title: Treatment of Prolonged Uterine Bleeding of Etonogestrel (ENG)-Releasing Implant Using Norethisterone (NET)-Only Pill: a Randomized Controlled Trial
Brief Title: Treatment of Prolonged Uterine Bleeding of Etonogestrel (ENG)-Releasing Implant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Organon (Industry)
Responsible Party: Principal Investigator, Carolina Sales Vieira, Professor, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3.396.056
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Breakthrough Bleeding
Keywords: norethisterone; uterine bleeding; progestogen-only contraceptives; etonogestrel-releasing implant
MeSH Terms: conditions — Metrorrhagia; Uterine Hemorrhage | interventions — Norethindrone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Norethisterone 10mg/day (Experimental): NET-only pill (Norethisterone, Primolut-Nor®), 10 mg/day, 1 pill per day until 2 consecutive days without bleeding/spotting (maximum use of 1 box of Primolut-Nor® per bleeding episode)
  Interventions: Drug: Norethisterone 10mg/day
- Placebo (Placebo Comparator): Identically appearing placebo to Primolut-Nor®, 1 pill per day until 2 consecutive days without bleeding/spotting (maximum use of 1 box of Placebo per bleeding episode)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Norethisterone 10mg/day — NET-only pill (Norethisterone, Primolut-Nor®), 10 mg/day, 1 pill per day until 2 consecutive days without bleeding/spotting
  Other Names: Primolut-Nor®, 10 mg/day, 1 pill per day
  Arms: Norethisterone 10mg/day
Drug: Placebo — Identically appearing placebo to Primolut-Nor®, 1 pill per day until 2 consecutive days without bleeding/spotting
  Arms: Placebo

SUMMARY:
Long-acting reversible contraceptives [LARC; copper-intrauterine devices (IUDs), the levonorgestrel-releasing intrauterine system (LNG-IUS) and subdermal implants] are the most effective reversible contraceptives available. A common side effect of these methods is changes in menstrual bleeding. Dissatisfaction with unpredictable bleeding is the main reason for early discontinuation of LARC methods.

The mechanism of unpredictable bleeding is unknown; it is likely related to the progestogen dilating superficial veins and capillaries, which are fragile and susceptible to focal bleeding. Other potential influences include changes in structural support of the endometrium, altered matrix metalloproteinase activity, and changes in endometrial perfusion and hemostasis. Local genetic alterations of the hormonal receptors of endometrium can also play a role in the etiology of the unpredictable bleeding experienced by some women.

Regarding etonogestrel (ENG)-releasing implant, some evidences suggest that the use of mefenamic acid, mifepristone with estradiol or doxycycline, or doxycycline alone can temporally stop the bleeding; however, all these therapies cannot avert the recurrence of the bleeding. Recently, a randomized clinical trial (RCT) evaluated the effectiveness of a short-term use of combined oral contraceptive (COC) in stopping bleeding episodes and preventing bleeding recurrence. The authors found that bothersome bleeding in ENG-implant users stopped within 14-day of COC treatment, but bleeding most often resumes within 10 days of treatment cessation.

Although COC can stop the bleeding, it is not known which component of the COC is responsible for this effect. There is evidence suggesting that estrogen alone is not effective in stopping the bleeding of progestogen-only contraceptives or a high dose of ethinyl estradiol is needed to obtain this effect. Furthermore, the recurrence of the bleeding shown with the COC use could be explained by the interruption of the estrogen. For this reason, our hypothesis is that a progestogen-only pill could be superior to placebo in stopping the bleeding associated with the ENG-implant use as well as being superior to placebo in recurrence of bleeding after discontinuation of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* To be an etonogestrel-releasing implant user for at least 40 days with a current bleeding/spotting episode of at least 7 consecutive days;
* Age between 18-40 years old;
* To have a mobile phone.

Exclusion Criteria:

* Body mass index (BMI; kg/m2) ≥ 35;
* Pregnancy;
* To have a positive chlamydia test;
* To be unable or unwilling to swallow pills;
* To have a medical condition deemed severe by a physician investigator;
* To be in use of a hepatic enzyme inducing medication;
* To be in use of anticoagulant drug;
* To have findings on speculum examination indicating an anatomic source of bleeding (e.g., polyp, cervicitis);
* To be in the first 6 months of delivery;
* To be on a concurrent hormonal contraceptive, depot medroxyprogesterone acetate (DMPA) interruption ≤ 6 months;
* To be illiterate;
* To be in use of any drug to stop the bleeding associated with etonogestrel implant ≤ 15 days.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Percentage of women who will stop the prolonged uterine bleeding after 7 days of medication use. | 7 days
  We will measure the percentage of women will stop the uterine bleeding after 7 days of norethisterone or placebo use. Participants will report their bleeding and/or spotting through text messages and daily diary.

SECONDARY OUTCOMES:
Number of days of medication use until interruption of uterine bleeding episode | 30 days
  We will analyze the mean (95%CI) number of days of placebo and norethisterone use until interruption of uterine bleeding episode. Participants will report their bleeding and/or spotting through text messages and daily diary. Women will use it until being 2 days without uterine bleeding/spotting or until the end of the box if the bleeding does not stop earlier.
Percentage of women who will stop the prolonged uterine bleeding after 14 days of medication use. | 14 days
  We will measure the percentage of women will stop the uterine bleeding after 14 days of norethisterone or placebo use. Participants will report their bleeding and/or spotting through text messages and daily diary.
The interval (number of days) to the recurrence of uterine bleeding after discontinuation of the first treatment cycle. | 6 months
  Participants will report their bleeding and/or spotting through text messages and daily diary. Women will use the randomized drug until being 2 days without uterine bleeding/spotting or until the end of the box if the bleeding does not stop earlier. We will assess the mean number of days (95%CI) until a new bleeding episode occur.
Bleeding patterns within 6 months after the end of the first treatment cycle | 6 months
  We will summarize the bleeding patterns according to the World Health Organization terminology. Participants will report their bleeding and/or spotting through text messages and daily diary.
Percentage of women who will need to repeat the treatment in order to stop the uterine bleeding (none vs. 1-2 times vs. 3 times) | 6 months
  Women can repeat the same treatment 3 times in the following 6 months of follow-up in case of a new bleeding/spotting episode of at least 7 consecutive days. Participants will report their bleeding and/or spotting through text messages and daily diary. Women will the randomized drug until being 2 days without uterine bleeding/spotting or until the end of the box if the bleeding does not stop earlier. We will assess the percentage of women who will need to repeat the treatment in order to stop new uterine bleeding episodes (none vs. 1-2 times vs. 3 times)
Relation between plasmatic levels of etonogestrel and bleeding patterns at baseline and at 7 days of randomized drug use | 7 days
  We will evaluate the etonogestrel level using Ultra Pressure Liquid Chromatography and will perform a multiple analysis to see if unfavorable bleeding patterns are related with etonogestrel levels.
Treatment failure | 30 days
  Percentage of treatment failure in each study arm. Treatment failure is defined by the maintenance of the bleeding episode after 30 days of continuous drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina S Vieira, PhD, MD, Study Chair — Professor
Locations (2):
- Brazil (2):
  - Unidade de Pesquisa Clínica do Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo
  - UNIFESP, São Paulo, São Paulo